CLINICAL TRIAL: NCT04571983
Title: Influence of Reliance on Historical Blood Eosinophil Counts on ICS Prescribing by GOLD 2019 Thresholds in COPD
Acronym: BECCOPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 285200
Record Dates: First submitted 2020-08-12; First posted 2020-10-01 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Eosinophil counts - comparing historical with stable state — Comparing historical blood eosinophil counts over 24 months to stable state eosinophil count.

SUMMARY:
Blood eosinophils are a type of white blood cell that helps fight infection. They have a number of different functions but are primarily involved in numerous inflammatory processes. They are recruited from the blood into sites of inflammation.

In patients with COPD, higher blood eosinophil count (BEC) predicts a greater reduction in moderate and severe exacerbations in response to inhaled corticosteroid (ICS) therapy. The Global Initiative for Chronic Obstructive Lung Disease strategy (GOLD 2019) recommends the use of BEC to guide ICS therapy and states that eosinophil levels above 300 cells/μL can help identify responders, guiding initial dual therapy, with "little or no effect at a BEC < 100 cells/μL". The National Institute for Health and Care Excellence (NICE) COPD 2018 guideline states that a higher BEC is associated with ICS response, but does not specify a threshold. Earlier research studies have suggested that at lower levels of BEC the harm of ICS due to pneumonia is greater than the benefit of severe exacerbation reduction.

Patients with COPD can have "flare ups" of their disease known as exacerbations. Blood eosinophils play a critical role in assessing severity of these exacerbations and guiding management. The association between BEC and reduction in exacerbation frequency is based on BEC measured when the patient is clinically stable. Transient low eosinophil count (eosinopenia with BEC < 50 cells/μL) during severe exacerbation is extremely common. In the Dyspnoea, Eosinopenia, Consolidation, Acidaemia and atrial Fibrillation (DECAF) score derivation and validation studies combined, eosinopenia was present on admission in 1,340 of 2,645 severe exacerbations of COPD (ECOPD) and is associated with longer length of stay, higher in-hospital and one year mortality. Although eosinophilic COPD exacerbations occur, overall BEC during moderate or severe exacerbation is lower than stable state.

In ECOPD managed in critical care low BEC is associated with higher rate of septic shock and mortality. BEC are also suppressed during other acute illnesses, notably sepsis. Failure to recognise that BEC are often suppressed during acute illness compared to stable state may lead to ICS therapy being inappropriately withheld. The effect of exacerbation and other acute illnesses on eosinophils is under-appreciated. Both NICE and GOLD guidelines fail to mention whether BEC should be prospectively measured when patients are stable (reflecting RCT evidence), or if reliance on historical values is acceptable.

In routine practice some clinicians rely on previous BECs to avoid a delay in treatment decisions. A number of these historical counts will have been taken during illness, underestimating the patients' stable-state BEC. Conversely, COPD is associated with other medical conditions, and BEC may be requested for reasons other than acute illness. Using the highest BEC from multiple measures in the previous 24 months may therefore better agree with stable state counts.

The primary aim of this trial is to assess the reliability of using BEC over the preceding 24 months to assess COPD eosinophil phenotype at both GOLD thresholds. The primary outcome will be based on using the highest of at least three BEC. Secondary outcomes include a) the level of agreement between baseline stable state BEC and both mean and the highest BEC over the preceding 24 months, b) the influence of the number of BEC measures available and c) the effect of limiting the time frame from 24 months to the previous 12 months.

BEC is associated with disease severity, providing further evidence that COPD eosinophil phenotype may change over time. As an exploratory analysis, periods of sustained change in eosinophil phenotype will be sought, and the relationship between eosinophil phenotype and patient characteristics and certain medication will be assessed.

The investigators will also assess the relations between the dependent variables stable state absolute eosinophil and basophil counts and both eosinophil to basophil and neutrophil to lymphocyte ratios and the following clinical outcomes: a) moderate and severe exacerbations and b) mortality. Some of these variables have previously been shown to be related to disease severity and mortality.

DETAILED DESCRIPTION:
In patients with COPD, higher blood eosinophil count (BEC) predicts a greater reduction in moderate and severe exacerbations in response to inhaled corticosteroid (ICS) therapy. The Global Initiative for Chronic Obstructive Lung Disease strategy (GOLD 2019) recommends the use of BEC to guide ICS therapy and states that eosinophil levels above 300 cells/μL can help identify responders, guiding initial dual therapy, with "little or no effect at a BEC < 100 cells/μL". The National Institute for Health and Care Excellence (NICE) COPD 2018 guideline states that a higher BEC is associated with ICS response, but does not specify a threshold. An earlier post hoc risk-benefit analysis suggested that at lower levels of BEC the harm of ICS due to pneumonia is greater than the benefit of severe exacerbation reduction.

The association between BEC and reduction in exacerbation frequency is based on BEC measured when the patient is clinically stable. Transient eosinopenia (BEC < 50 cells/μL) during severe exacerbation is extremely common. In the Dyspnoea, Eosinopenia, Consolidation, Acidaemia and atrial Fibrillation (DECAF) score derivation and validation studies combined, eosinopenia was present on admission in 1,340 of 2,645 severe exacerbations of COPD (ECOPD) and is associated with longer length of stay (DECAF combined cohorts: median difference 1 day, p<0.001 unpublished data), and higher in-hospital and one year mortality. Although eosinophilic COPD exacerbations occur, overall BEC during moderate or severe exacerbation is lower than stable state. In ECOPD managed in critical care low BEC is associated with higher Acute Physiology, Age, Chronic Health Evaluation II (APACHE II) scores, rate of septic shock and mortality. BEC are also suppressed during other acute illnesses, notably sepsis. Failure to recognise that BEC are often suppressed during acute illness compared to stable state may lead to ICS therapy being inappropriately withheld. Regrettably, whilst the effect of eosinophils on exacerbation is well recognised, the effect of exacerbation and other acute illnesses on eosinophils is under- appreciated. Both NICE and GOLD fail to mention whether BEC should be prospectively measured when patients are stable (reflecting RCT evidence), or if reliance on historical values is acceptable.

In routine practice some clinicians rely on previous BECs to avoid a delay in treatment decisions. A number of these historical counts will have been taken during illness, underestimating the patients' stable-state BEC. Conversely, COPD is associated with multimorbidity, and BEC may be requested for reasons other than acute illness. Using the highest BEC from multiple measures in the previous 24 months may therefore better agree with stable state counts.

The primary aim of this trial is to assess the reliability of using BEC over the preceding 24 months to assess COPD eosinophil phenotype at both GOLD thresholds. The primary outcome will be based on using the highest of at least three BEC. Secondary outcomes include a) the level of agreement between baseline stable state BEC and both mean and the highest BEC over the preceding 24 months, b) the influence of the number of BEC measures available and c) the effect of limiting the time frame from 24 months to the previous 12 months.

Whilst BEC is relatively stable over weeks and months, agreement wanes over longer timeframes. BEC is also associated with disease severity, providing further evidence that COPD eosinophil phenotype may change over time. As an exploratory analysis, periods of sustained change in eosinophil phenotype will be sought, and the relationship between eosinophil phenotype and patient characteristics and medication (including prophylactic azithromycin) will be assessed. Recent work suggests that a low Eosinophil to Basophil ratio predicts exacerbation risk and mortality, whilst a high neutrophil to lymphocyte ratio is related to disease severity, exacerbations and mortality.

The investigators will also assess the relations between the dependent variables stable state absolute eosinophil and basophil counts and both eosinophil to basophil and neutrophil to lymphocyte ratios and the following clinical outcomes: a) moderate and severe exacerbations and b) mortality.

Importance to the NHS

1. This study will assess the variation in BEC measured during both stable state and acute illness in patients with COPD. The investigators anticipate that the results will help prevent inappropriate denial of ICS therapy due to reliance on BEC sampled when a patient is unwell.

   Both NICE COPD guidelines and the GOLD strategy statement appropriately recommend that BEC should help direct ICS therapy in COPD, but fail to emphasise that the evidence supporting this advice is based solely on BEC measured when the patient is stable. BEC are suppressed during many acute illnesses, including severe exacerbations of COPD, and it is during these episodes that blood tests are most likely to taken. Reliance on BEC sampled during such episodes may lead to inappropriate denial of ICS therapy and increased risk of moderate and severe ECOPD.
2. This study will determine whether the highest of at least three BEC measured over the preceding 24 months provides an acceptable level of agreement with stable state BEC in terms of ICS treatment choice. In a sensitivity analysis, the investigators will assess the influence of using mean rather than highest BEC, the number of BEC available, and timeframe on this outcome.

In the world of realistic medicine, ensuring a patient attends their GP practice or hospital clinic for measurement of BEC when they are stable, and then returns when the result is available before a treatment decision is made is unlikely to be achieved in most cases. However multiple previous BEC are often available, and some are likely to have been measured during recovery or taken at other times when the patient was stable. The clinical systems used in primary and secondary care allow all previous BEC available for a patient to be collated and displayed on screen simply by clicking on a single eosinophil measurement. The outcome of this study will inform clinicians of the level of certainty several historical BEC provide in regard to ICS treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Physician confirmed COPD.
2. Age 35 or older.
3. Current or former smoker with 10+ pack years smoking history.
4. FEV1 <80% with FEV1/(F)VC < 0.7.
5. Three or more blood eosinophil counts performed within the last 24 months.
6. Clinically stable at the time of the baseline assessment, with no exacerbations of COPD or oral prednisolone therapy within the last 4 weeks.*
7. Capacity to give informed consent to participate.

   * The baseline assessment can be rescheduled for patients who do not meet the clinical stability criteria, provided they satisfy all other selection criteria.

Exclusion Criteria:

1. Maintenance oral prednisolone or other systemic steroids, anti-interleukin-5 therapy or other medication known to suppress eosinophils.
2. Active malignancy.
3. Investigator confirmed history of asthma.†
4. Parasitic infection, systemic fungal infection (excluding infection limited to nails or skin), eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome or other conditions associated with a high eosinophil count.‡
5. Drug or alcohol problems which in the view of the primary investigatory may compromise the conduct and completion of the study.

   * Asthma and COPD may co-exist, but both conditions are also commonly misdiagnosed. Only patients who in the view of the investigator have asthma, and therefore should receive ICS therapy, will be excluded.

     * Patients with atopic conditions such as allergic rhinitis, allergic conjunctivitis and eczema will be eligible.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified within primary and secondary care. The lead centre has a research database of patients who have participated in previous trials, and both units have strong links with primary care. Recruitment will be supported by engaging primary care Participant Identification Centre (PIC) sites. Patients will also be identified following attendance at clinic or pulmonary rehabilitation, and following admission with an exacerbation of COPD. Those that meet selection criteria, including confirmation of clinical stability on study entry, will be invited to consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The agreement between the highest BEC within the previous 24 months and baseline stable-state BEC following dichotomisation into < 300 cells/μL and ≥ 300 cells/μL. | historical eosinophil counts previous 24 months: prospective follow up for 3 months

SECONDARY OUTCOMES:
The agreement between the highest BEC within the previous 24 months and baseline stable- state BEC following dichotomisation into < 100 cells/μL and ≥ 100 cells/μL. | historical eosinophil counts previous 24 months: prospective follow up for 3 months
Comparison of agreement between a) the highest BEC within the previous 24 months and baseline stable-state BEC, and b) baseline and three month stable state BEC. This will be performed at both thresholds (100 and 300 cells/μL). | historical eosinophil counts previous 24 months: prospective follow up for 3 months
Sensitivity analyses: a) the influence of using the mean rather than the highest BEC within the previous 24 months on agreement with baseline stable-state BEC; b) influence of number of available BEC measures over last 24 months on the level of agreement | historical eosinophil counts previous 24 months: prospective follow up for 3 months
The agreement between both a) the highest BEC and b) the mean BEC within the previous 24 months and baseline stable-state using continuous data. | historical eosinophil counts previous 24 months: prospective follow up for 3 months

OTHER OUTCOMES:
The rate of moderate and severe exacerbations will be compared with blood eosinophil count, both as a continuous measure and categorised by the GOLD 2019 treatment thresholds (BEC: 0-99; 100-299; 300+ cells/µL). | historical eosinophil counts previous 24 months: prospective follow up for 3 months
Non-elective hospital admissions over the 36 month study period will be identified and categorised by primary diagnosis. Admission BEC will be reported, with and without adjustment for oral glucocorticoid therapy. | historical eosinophil counts previous 24 months: prospective follow up for 3 months
An initial exploratory analysis will investigate changes in eosinophil count between patients at baseline and averaged over the follow up period. We will also look at changes over time across all patients, and the factors influencing this. | historical eosinophil counts previous 24 months: prospective follow up for 3 months
  The final part of the analysis will be a mixed model accounting for both within and between patient factors and their influence on each of the outcomes. Key covariates of interest will include a) FeNO, b) smoking status (current and ex-smokers), c) age, d) FEV1, e) azithromycin therapy
Association between the dependent variables: a) baseline eosinophil and basophil counts, b) eosinophil to basophil ratio, and c) neutrophil to lymphocyte ratio and the clinical outcomes: a) rate of moderate and severe exacerbations and b) mortality. | historical eosinophil counts previous 24 months: prospective follow up for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bourke, MBCHb, PhD, Principal Investigator — Northumbria Healthcare NHS Foundation Trust
Locations (1):
- North Tyneside General Hospital, North Shields, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be available for the primary research team